CLINICAL TRIAL: NCT06975241
Title: Determining Contribution of Sex and Genetics to DHA Synthesis Rates Over 12 Weeks of EPA Supplementation in Healthy Individuals
Brief Title: Observing Metabolism of EPA With Consideration of Genetics And Sex
Acronym: OMEGA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Adam Metherel, Assistant Professor, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 00048186
Record Dates: First submitted 2025-04-29; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Healthy; Omega 3; Metabolism, Lipids
Keywords: eicosapentaenoic acid; omega-3 polyunsaturated fatty acids; lipid metabolism; healthy adults; docosahexaenoic acid; single nucleotide polymorphism; elongation of very long-chain 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EPA Supplementation (Experimental): 32 males and 32 females will be enrolled in the EPA supplementation arm, with an equal number of GA+GG and AA genotypes (rs953413 SNP) among males and females.
  Interventions: Dietary Supplement: EPA 2.4g/day

INTERVENTIONS:
Dietary Supplement: EPA 2.4g/day — EPA from fish oil will be supplemented to an equal number of males and females for 12 weeks.

SUMMARY:
The goal of this clinical study is to learn how fast EPA is converted to other molecules, including DHA, with consideration of biological sex and genetics in healthy humans.

The main questions it aims to answer are:

* How fast is EPA converted to DHA in blood, and is the conversion rate affected by sex and a specific genotype we previously identified?
* How do sex and the specific genotypes affect blood DHA levels and other products of DHA in response to dietary EPA?
* How fast does dietary EPA replace blood EPA and other omega-3 fatty acids, and is the rate affected by sex and genotype?

Participants will be asked to take EPA supplements for 12 weeks and provide a series of venous blood samples over the study duration.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5- 30 kg/m2
* healthy

Exclusion Criteria:

* High consumption of n-3 PUFA, including ≥ 2 servings of fish/seafood or EPA/DHA-enriched foods per week
* Consumption of any supplements containing ALA/EPA/DHA currently or within the previous 6 months
* Allergies to any component of the study supplement (fish, gelatin etc.)
* BMI <18.5 kg/m² or >30 kg/m²
* Women who are pregnant, breastfeeding or planning on becoming pregnant
* Diagnosis with chronic or communicable diseases
* Prescription of chronic pharmacological medications (except for oral contraceptives)
* High blood pressure (systolic or diastolic blood pressure above 130 or 80mmHg, respectively)
* Hypertriglyceridemia (serum > or = 1.69 mmol/l)
* Hypercholesterolemia (serum LDL-C > or =5 mmol/l)
* Anticipated changes in lifestyle within the next 4 months
* Smoking
* Heavy alcohol use (>3 drinks/day)
* Major surgery in the last six months

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Plasma DHA synthesis/turnover rates | Day 0, 3, 7, 14, 28, 56, 84
  Plasma DHA synthesis/turnover rates (nmol/mL/day) by sex and rs953413 ELOVL2 polymorphism will be determined. DHA synthesis/turnover rates will be calculated from frequent sampling of plasma DHA levels and carbon-13 isotope signatures of DHA (δ13C-DHA) over 12 weeks.

SECONDARY OUTCOMES:
Changes in plasma DHA concentrations (nmol/ml) | Baseline and 12 weeks
  Changes in plasma DHA concentrations by sex and rs953413 ELOVL2 polymorphism will be determined.
Plasma EPA turnover rates (nmol/ml/day) | Day 0, 3, 7, 14, 28, 56, 84
  Plasma EPA turnover rates (nmol/mL/day) by sex and rs953413 ELOVL2 polymorphism will be determined. EPA turnover rates will be calculated from frequent sampling of plasma EPA levels and carbon-13 isotope signatures of EPA (δ13C-EPA) over 12 weeks.
Plasma DPAn-3 synthesis/turnover rates (nmol/ml/day) | Day 0, 3, 7, 14, 28, 56, 84
  Plasma DPAn-3 synthesis/turnover rates (nmol/mL/day) by sex and rs953413 ELOVL2 polymorphism will be determined. DPAn-3 synthesis/turnover rates will be calculated from frequent sampling of plasma DPAn-3 levels and carbon-13 isotope signatures of DPAn-3 (δ13C-DPAn-3) over 12 weeks.
Changes in PUFA derived eicosanoid/docosanoid levels | Baseline, 4 weeks and 12 weeks
  Changes in n-3 and n-6 PUFA derived eicosanoid/docosanoid levels by sex and rs953413 ELOVL2 polymorphism will be investigated.
Plasma half-lives of EPA and downstream n-3 PUFAs | Over 12 weeks
  Plasma half-lives of EPA and downstream n-3 PUFAs (in days) will be determined with the consideration of sex and rs953413 ELOVL2 polymorphism.

OTHER OUTCOMES:
Changes in plasma and erythrocyte levels of all fatty acids | Baseline and 12 weeks
  Changes in plasma and erythrocyte levels of all fatty acids by sex and rs953413 ELOVL2 polymorphism will be investigated.
Changes in plasma δ13C signature of all fatty acids | Baseline and 12 weeks
  Changes in plasma δ13C signature (mUr) of all fatty acids with consideration of sex and rs953413 ELOVL2 polymorphism will be investigated.
Changes in plasma oxylipin levels | Baseline, 4 weeks and 12 weeks
  Changes in other oxylipin levels with consideration of sex and rs953413 ELOVL2 polymorphism will be investigated.
Synthesis/turnover rates of EPA and downstream n-3 PUFAs (nmol/ml/day) according to sex and additional genetic polymorphisms | Day 0, 3, 7, 14, 28, 56, 84
  Plasma synthesis/turnover rates of EPA and downstream n-3 PUFAs will be investigated according to the effect of sex and additional genetic polymorphisms (in the FADS gene cluster, ELOVL2, ELOVL5 and ACOX).
Change in levels of EPA and downstream n-3 PUFAs according to sex and additional genetic polymorphisms | Baseline and 12 weeks
  Change from baseline in levels of EPA and downstream n-3 PUFAs will be investigated according to sex and additional genetic polymorphisms (in the FADS gene cluster, ELOVL2, ELOVL5 and ACOX)
Plasma synthesis/turnover rates of EPA and downstream n-3 PUFAs (nmol/ml/day) according to blood circulating nutrients and genetic polymorphisms | Day 0, 3, 7, 14, 28, 56, 84
  Plasma synthesis/turnover rates of EPA and downstream n-3 PUFAs (nmol/ml/day) will be investigated according to the interaction of blood circulating nutrients (vitamin B6, nicotinic acid, zinc, iron, magnesium, calcium) and genetic polymorphisms (in FADS gene cluster, ELOVL2 and ELOVL5).
Change in plasma levels of EPA and downstream n-3 PUFAs according to blood circulating nutrients and genetic polymorphisms | Baseline and 12 weeks
  Change from baseline in plasma levels of EPA and downstream n-3 PUFAs will be investigated according to the interaction of blood circulating nutrients (vitamin B6, nicotinic acid, zinc, iron, magnesium, calcium) and genetic polymorphisms (in FADS gene cluster, ELOVL2 and ELOVL5).
Adherence | Baseline and 12 weeks
  Adherence to supplementation will be assessed by capsule count, change in plasma EPA levels and change in δ13C signature of EPA
Changes in blood lipid profile | Baseline and 12 weeks
  Changes in lipid profile including triglycerides, LDL, HDL, total cholesterol, and non-HDL (mmol/L) with consideration of sex and rs953413 ELOVL2 polymorphism will be investigated.
Changes in office blood pressure (mmHg) | Day 0, 14, 28, 56, 84
  Changes in office systolic and diastolic blood pressure (mmHg) with consideration of sex and rs953413 ELOVL2 polymorphism will be investigated.
Changes in heart rate (bpm) | Day 0, 14, 28, 56, 84
  Changes in heart rate (bpm) with consideration of sex and rs953413 ELOVL2 polymorphism will be investigated.
Symptoms Diary | Throughout 12 weeks
  To monitor safety throughout the study, participants will report any unusual symptoms in a symptoms diary. The symptom will be described, along with the date of occurrence and the severity of the symptom on a scale of 1 (low) to 7 (high).
Dietary intake | Day 0, 28, 56, 84
  Dietary intake in males and females will be assessed by estimated 3 day food record at baseline and days 28, 56 and 84.
Body mass index (kg/m²) | Day 0, 28, 56, 84
  BMI (kg/m²) will be calculated by the measure of height (metres) and weight (kilograms) throughout the study.
Body fat percentage | Day 0, 28, 56, 84
  Body fat percentage as measured by bioelectrical impedance will be determined.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition and Risk Factor Modification Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
IPD that resulted in a publication will be shared in a de-identified/anonymized format.
Time Frame: Beginning 1 year after publication of the data with no end date.
Access Criteria: IPD will be accessible through University of Toronto dataverse (https://borealisdata.ca/dataverse/toronto). The metadata record will be public but access to the dataset will be restricted. Users will need to request access to view and download the dataset.